CLINICAL TRIAL: NCT01729819
Title: A Multi-centre, Double-blind, Randomised Trial Investigating the Efficacy and Safety of a Combination Therapy, Desmopressin and Tolterodine, for Treatment of Overactive Bladder With Nocturia in Women
Brief Title: Interventional Clinical Trial in Patients in Overactive Bladder With Nocturia in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000085
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination (Experimental): Tolterodine tartrate extended release capsules + Desmopressin orally disintegrating tablets
  Interventions: Drug: Tolterodine tartrate extended release capsules; Drug: Desmopressin orally disintegrating tablets
- Tolterodine (Active Comparator): Tolterodine tartrate extended release capsules + Placebo orally disintegrating tablets
  Interventions: Drug: Tolterodine tartrate extended release capsules; Drug: Placebo orally disintegrating tablets

INTERVENTIONS:
Drug: Tolterodine tartrate extended release capsules
Drug: Desmopressin orally disintegrating tablets
  Arms: Combination
Drug: Placebo orally disintegrating tablets
  Arms: Tolterodine

SUMMARY:
The purpose of the trial is to investigate the efficacy of combining tolterodine and desmopressin compared with tolterodine monotherapy in the treatment of women with overactive bladder with nocturia in terms of reduction of nocturnal voids during 3 months of treatment

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to performance of any trial-related activity
* Female sex, at least 18 years of age (at the time of written consent)
* Nocturia and overactive bladder symptoms present for ≥6 months prior to trial entry (patient-reported)
* At least 2 nocturnal voids each night as documented in 2 diary periods during the screening. A mean of at least 8 daytime voids per day over 3 days with a minimum of at least 6 daytime voids each day as documented in 2 diary periods during the screening. At least 1 urgency episode each 24 hours as documented in 2 diary periods during the screening. Each diary period consists of 3 consecutive days, with at least 14 days between each period.

Exclusion Criteria:

* Evidence of severe voiding dysfunction defined as:

More than 10 nocturnal voids per 24 hours as documented on any of the days in both diary periods during screening.

More than 20 daytime voids per 24 hours as documented on any of the days in both diary periods during screening.

* Genito-urinary tract pathology that can in the investigator's opinion be responsible for urgency or urinary incontinence e.g., symptomatic or recurrent urinary tract infections, interstitial cystitis, bladder related pain, or stone in the bladder and urethra causing symptoms
* Current or a history within 5 years of lower urologic malignancies (e.g., bladder cancer), lower urinary tract surgery, previous pelvic irradiation, or severe neurological disease affecting bladder function or muscle strength (e.g., multiple sclerosis, Parkinson's disease, spinal cord injury, spina bifida)
* Symptoms of severe stress urinary incontinence in the opinion of the investigator
* Urinary retention or a post void residual volume in excess of 150 mL as confirmed by bladder ultrasound performed after suspicion of urinary retention
* Habitual or psychogenic polydipsia (fluid intake resulting in a urine production exceeding 40 mL/kg/24 hours) or a mean volume voided per void of 350 mL or more during one or more 24-hour periods as assessed by the screening diaries
* Central or nephrogenic diabetes insipidus
* Syndrome of inappropriate antidiuretic hormone (SIADH)
* Gastric retention
* Myasthenia gravis
* Uncontrolled narrow-angle glaucoma
* Suspicion or evidence of cardiac failure
* Uncontrolled and clinically relevant (in the judgement of the investigator) hypertension or diabetes mellitus
* History and/or current treatment of obstructive sleep apnoea
* Hyponatraemia:Serum sodium level must not be below 135 mmol/L
* Evidence of potential renal impairment:Serum creatinine must be within normal laboratory reference intervals AND estimated glomerular filtration rate must be more than or equal to 50 mL/min
* Hepatic and/or biliary diseases: Aspartate aminotransferase and/or alanine aminotransferase levels must not be more than twice the upper limit of normal range. Total bilirubin level must not be more than 1.5 mg/dL
* Pregnancy, breastfeeding, or a plan to become pregnant during the period of the trial. Women of reproductive age must have documentation of a reliable method of contraception. All pre- and perimenopausal women have to perform pregnancy tests. Amenorrhea of more than 12 months duration based on the reported date of the last menstrual period is sufficient documentation of post-menopausal status and does not require a pregnancy test
* Known alcohol or substance abuse; work or lifestyle that may interfere with regular night-time sleep e.g., shift workers; or any other medical condition, laboratory abnormality, psychiatric condition, mental incapacity, illiteracy or language barrier which, in the judgement of the investigator, would impair participation in the trial
* Known or suspected hypersensitivity to any active ingredient or excipients in the investigational medicinal products used in the trial
* Previous participation in any desmopressin trial within the last 5 years
* Use of any prohibited therapy, as defined in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (24):
- United States (24):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Lynn Institute of The Ozarks, Little Rock, Arkansas
  - Moez Khorsandi, DO, Los Angeles, California
  - Urology Group of Southern California, Los Angeles, California
  - Riverside Clinical Research, Edgewater, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northshore Center for Gastroenterology, Evanston, Illinois
  - Remedica, LLC, Rochester, Michigan
  - The Urological Institute of Northeastern New York, Albany, New York
  - Premier Medical Group of the Hudson Valley, P.C., Poughkeepsie, New York
  - Parkhurst Research Organization, LLC, Bethany, Oklahoma
  - Philadelphia Clinical Research, LLC, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Research Across America, Dallas, Texas
  - Advances in Health, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Radiant Research, San Antonio, Texas
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-centre trial conducted in the US. A total of 33 sites were initiated in this trial, and of these eligible patients from 20 sites were randomised to a treatment. The first patient first visit was on 28 January 2013. The last patient last visit was on 19 November 2014.
Pre-assignment Details: The trial was initiated with a screening period of 3-4 weeks between Visits 1 and 2a, where no investigational medicinal product was taken. Patients who were on a prohibited medication and needed a wash-out period of 1-2 weeks initiated the trial at Visit 0. Eligible patients were randomised to one of the two treatment groups at Visit 2a.
Groups:
- Combination: Tolterodine tartrate extended release capsules (4 mg) + Desmopressin orally disintegrating tablets (25 μg)
  Tolterodine tartrate extended release capsules
  Desmopressin orally disintegrating tablets
- Tolterodine: Tolterodine tartrate extended release capsules (4 mg) + Placebo orally disintegrating tablets
  Tolterodine tartrate extended release capsules
  Placebo orally disintegrating tablets
Period: Overall Study
Arm/Group | Combination | Tolterodine
Started (The ITT comprised of all randomised patients (49 in combination group and 57 in tolterodine group)) | 49 | 57
Completed | 43 | 50
Not Completed | 6 | 7
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other reason | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised of all randomised and exposed subjects with at least one efficacy assessment after treatment initiation.The FAS comprised of 97 subjects (45 in the combination group and 52 in the tolterodine group). All analyses were done based on the FAS.
Groups:
- Combination: Tolterodine tartrate extended release capsules (4 mg) + Desmopressin orally disintegrating tablets (25 µg)
  Tolterodine tartrate extended release capsules
  Desmopressin orally disintegrating tablets
- Tolterodine: Tolterodine tartrate extended release capsules (4 mg)+ Placebo orally disintegrating tablets
  Tolterodine tartrate extended release capsules
  Placebo orally disintegrating tablets
- Total: Total of all reporting groups
Arm/Group | Combination | Tolterodine | Total
Number analyzed (Participants) | 45 | 52 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (12.6) | 51.8 (10.3) | 53.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 52 | 97
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 33 | 42 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 35 | 38 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mean Number of Nocturnal Voids [Mean (Standard Deviation); unit: Voids] | 3.38 (0.97) | 3.11 (1.06) | 3.24 (1.02)
Mean Number of Day time Voids [Mean (Standard Deviation); unit: Voids] | 9.69 (1.35) | 10.1 (1.97) | 9.91 (1.71)
Mean Nocturnal Urine Volume [Mean (Standard Deviation); unit: mL] | 546 (281) | 537 (278) | 541 (278)
Mean Time to First Nocturnal Void [Mean (Standard Deviation); unit: Minutes] | 125 (44.6) | 143 (56.1) | 135 (51.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Nocturnal Voids From Baseline
Description: A nocturnal void was defined as a void occurring at least 5 minutes after going to bed, but before getting up the next morning. The mean estimate was the average over 3 consecutive 24-hour periods prior to the respective visit as captured in the voiding and sleep diary.
Time Frame: Baseline to 3 months of treatment
Population: The FAS comprised of all randomised and exposed subjects with at least one efficacy assessment after treatment initiation. The FAS comprised of 97 subjects (45 in the combination group and 52 in the tolterodine group).
Measure: Least Squares Mean (95% Confidence Interval); unit: Voids
Groups:
- Combination: Tolterodine tartrate extended release capsules (4 mg)+ Desmopressin orally disintegrating tablets (25 μg)
  Tolterodine tartrate extended release capsules
  Desmopressin orally disintegrating tablets
Arm/Group | Combination | Tolterodine
Number analyzed (Participants) | 45 | 52
Voids | -1.63 [-1.94 to -1.32] | -1.29 [-1.57 to -1.00]
Statistical Analysis 1: Comparison: Combination vs Tolterodine; Combination versus tolterodine (i.e. effect in combination group minus effect in tolterodine group) is presented. The trial was to be declared positive if a statistically significant (two-sided, p < 0.05) positive effect for combining tolterodine and desmopressin compared to tolterodine monotherapy on the primary endpoint had been demonstrated; Test type: Superiority — The change in mean nocturnal voids from baseline as the dependent variable, baseline mean nocturnal voids as a covariate, and treatments and visit (Month 1, Month 2, and Month 3) as factors, was considered for the analysis. Longitudinal analysis based on repeated measures using analysis of covariance with subject as random effect. Missing values post-baseline were not imputed; p = 0.112, ANCOVA; Change in mean nocturnal voids as the dependent variable and baseline mean nocturnal voids as a covariate, treatment and visit as factors; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.77 to 0.08] — Longitudinal analysis based on repeated measures using analysis of covariance with subject as random effect. The estimated value represents the contrast of combination - tolterodine

2. Secondary Outcome: Change in Mean Time to First Nocturnal Void From Baseline
Description: The time to first nocturnal void was defined as the time from going to bed with the intention of sleeping until first nocturnal void or until waking in the morning in the case there is no nocturnal void. The time to first void was calculated as the average over three consecutive 24-hour periods prior to the respective visits.
Time Frame: Baseline to 3 months of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Combination | Tolterodine
Number analyzed (Participants) | 45 | 52
Minutes | 118.19 [88.53 to 147.85] | 100.19 [72.67 to 127.72]
Statistical Analysis 1: Comparison: Combination vs Tolterodine; Combination versus tolterodine (i.e. effect in combination group minus effect in tolterodine group) is presented; Test type: Superiority; p = 0.385, ANCOVA; Change in mean time to first void as dependent variable and baseline mean time to first void as a covariate, and treatment and visit as factors; Mean Difference (Final Values) = 18, 95% CI 2-sided [-22.96 to 58.96] — The estimated value represents the contrast of combination - tolterodine

3. Secondary Outcome: Change in Mean Nocturnal Urine Volume From Baseline
Description: The mean nocturnal urine volume was derived from the three-day urine volume diary. The nocturnal volume was defined as the sum of the volumes for all nocturnal voids including the volume of the first morning void within 30 min of waking up in the morning.
Time Frame: Baseline to 3 months of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Combination | Tolterodine
Number analyzed (Participants) | 45 | 52
mL | -156.6 [-212.88 to -100.37] | -92.46 [-145.27 to -39.66]
Statistical Analysis 1: Comparison: Combination vs Tolterodine; Combination versus tolterodine (i.e. effect in combination group minus effect in tolterodine group) is presented; Test type: Superiority; p = 0.103, ANCOVA; Change in mean nocturnal volume as the dependent variable and baseline mean nocturnal volume as a covariate, and treatment and visit as factors; Mean Difference (Final Values) = -64.16, 95% CI 2-sided [-141.46 to 13.14] — The estimated value represents the contrast of combination - tolterodine

4. Secondary Outcome: Responder Status
Description: Responder status was defined as ≥33% decrease in the mean number of nocturnal void and at least one night with no voids out of the 3-day diary period.
Time Frame: Baseline to 3 months of treatment
Population: as for outcome 1
Measure: Number; unit: Proportion of responders
Arm/Group | Combination | Tolterodine
Number analyzed (Participants) | 45 | 52
Proportion of responders | 0.40 | 0.29
Statistical Analysis 1: Comparison: Combination vs Tolterodine; Combination versus tolterodine (i.e. odds of being responder in combination group versus odds of being responder in tolterodine group) is presented. The proportion of responders during three months of treatment was analysed (i.e. the odds ratio of the odds of being a responder) longitudinally using Generalised Estimating Equation (GEE) for a repeated logistic regression; Test type: Superiority; p = 0.352, Generalized Estimating Equation — 33% responder status as dependent variable, baseline mean nocturnal voids as covariate, treatment, and visit as factors; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.71 to 2.62]

5. Secondary Outcome: Onset of Effect as Seen in Change in Mean Number of Nocturnal Voids From Baseline for Each Visit During Three Months of Treatment
Description: as for outcome 1
Time Frame: Baseline to 3 months of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Voids
Groups:
- Treatment Difference (Combination-tolterodine): Change in mean number of nocturnal voids between combination (desmopressin [25 µg] + tolterodine [4 mg]) and tolterodine (4 mg) was estimated at month 1, month 2, month 3 and overall during the three months
Arm/Group | Treatment Difference (Combination-tolterodine)
Number analyzed (Participants) | 97
Voids
  Month 1 | -0.19 [-0.68 to 0.30]
  Month 2 | -0.44 [-0.95 to 0.06]
  Month 3 | -0.43 [-0.86 to 0.01]
  Overall (during the three months) | -0.35 [-0.78 to 0.08]
Statistical Analysis 1: Comparison: Treatment Difference (Combination-tolterodine); Treatment difference (Combination-tolterodine) at Month 1; Test type: Superiority — Estimated contrast (Combination - tolterodine) from longitudinal analysis including a treatment-by visit interaction term; p = 0.443, ANCOVA — Adjusted treatment difference (Combination-tolterodine) in mean number of nocturnal voids at Month 1
Statistical Analysis 2: Comparison: Treatment Difference (Combination-tolterodine); Treatment difference (Combination-tolterodine) at Month 2; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.086, ANCOVA — Adjusted treatment difference in mean number of nocturnal voids (Combination-tolterodine) at Month 2
Statistical Analysis 3: Comparison: Treatment Difference (Combination-tolterodine); Treatment difference (Combination-tolterodine) at Month 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.055, ANCOVA — Adjusted treatment difference (Combination-tolterodine) in mean number of nocturnal voids at Month 3
Statistical Analysis 4: Comparison: Treatment Difference (Combination-tolterodine); Treatment difference (Combination-tolterodine) for the duration of 3 months; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.106, ANCOVA — Adjusted treatment difference (Combination-tolterodine) in mean number of nocturnal voids for the duration of 3 months

6. Secondary Outcome: Change in the Impact on Sleep as Measured by the Sleep Rating Scales From Baseline
Description: An electronic diary was used in the trial to document the impact on sleep quality (sleep rating scales). The sleep rating scales included three questions that ranged from 0 (poor) to 10 (good). The average of each question for each visit was summarised and the change from baseline was analysed longitudinally during the three months of treatment.
Time Frame: Baseline to 3 months of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Combination | Tolterodine
Number analyzed (Participants) | 45 | 52
Score on scale
  From very tired to wide awake, how do you feel now | 1.76 [1.31 to 2.21] | 1.33 [0.91 to 1.76]
  Rate how refreshed you feel now | 1.81 [1.37 to 2.24] | 1.46 [1.06 to 1.87]
  Rate the quality of your sleep last night | 1.95 [1.52 to 2.39] | 1.67 [1.27 to 2.08]
Statistical Analysis 1: Comparison: Combination vs Tolterodine; Combination versus tolterodine (i.e. score on scale in combination group versus score on scale in tolterodine group) is presented.Statistical analysis for "from very tired to wide awake, how do you feel now"; Test type: Superiority; p = 0.178, ANCOVA; Quality of sleep rating score as dependent variable, baseline quality of sleep rating scale value as a covariate, and responder status as a factor; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.20 to 1.05] — Estimated contrast (Combination - tolterodine) from longitudinal analysis of covariance
Statistical Analysis 2: Comparison: Combination vs Tolterodine; Combination versus tolterodine (i.e. score on scale in combination group versus score on scale in tolterodine group) is presented. Statistical analysis for "Rate how refreshed you feel now"; Test type: Superiority; p = 0.257, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.26 to 0.94] — Estimated contrast (Combination - tolterodine) from longitudinal analysis of covariance
Statistical Analysis 3: Comparison: Combination vs Tolterodine; Combination versus tolterodine (i.e. score on scale in combination group versus score on scale in tolterodine group) is presented. Statistical analysis for "Rate the quality of your sleep last night"; Test type: Superiority — Quality of sleep rating score as dependent variable, baseline quality of sleep rating scale value as a covariate, and responder status as a factor; p = 0.360, ANCOVA; Longitudinal analysis of covariance on change from baseline with baseline as a covariate, and treatment and visit as factors; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.32 to 0.88] — Estimated contrast (Combination - tolterodine) from longitudinal analysis of covariance

ADVERSE EVENTS:
Time Frame: 3 months
Description: The safety analysis set included all patients who received at least one dose of IMP and had at least one safety assessment. The safety analysis set comprised of 103 patients (48 in the combination group and 55 in the tolterodine group).
Groups:
- Combination: Tolterodine tartrate extended release capsules + Desmopressin orally disintegrating tablets
  Tolterodine tartrate extended release capsules
  Desmopressin orally disintegrating tablets
- Tolterodine: Tolterodine tartrate extended release capsules + Placebo orally disintegrating tablets
  Tolterodine tartrate extended release capsules
  Placebo orally disintegrating tablets
Arm/Group | Combination | Tolterodine
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/55
Other Adverse Events (participants affected / at risk) | 3/48 | 9/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination (N=48) | Tolterodine (N=55)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the Sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the Sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow the Sponsor to seek patent protection of the invention.